CLINICAL TRIAL: NCT00307099
Title: Randomized, Multi-Center, Comparative Trial of Short-Course Empiric Antibiotic Therapy Versus Standard Antibiotic Therapy for Subjects With Pulmonary Infiltrates in the Intensive Care Unit (ICU): Impact on Antimicrobial Resistance, Superinfections, Length of ICU Stay and Hospitalization, and Mortality
Brief Title: Comparative Antibiotic Therapy for Subjects With Pulmonary Infiltrates in the ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-216; BAMSG 4-02
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2007-02

CONDITIONS: Bacterial Infection
Keywords: bacterial diseases
MeSH Terms: conditions — Bacterial Infections | interventions — Meropenem

ARMS (2):
- Meropenem (Experimental): Meropenem 1 gram intravenously every 8 hours for 3 days (9 doses), then an additional 5 days if the Clinical Pulmonary Infection Score is greater than 6.
  Interventions: Drug: Meropenem
- Standard antibiotic therapy (Active Comparator): Standard intravenous antibiotic therapy for a minimum of 8 days.
  Interventions: Drug: Standard antibiotic therapy

INTERVENTIONS:
Drug: Meropenem — Meropenem 1 gram intravenously every 8 hours for 3 days (9 doses), then an additional 5 days if the Clinical Pulmonary Infection Score is greater than 6.
  Arms: Meropenem
Drug: Standard antibiotic therapy — Standard intravenous antibiotic therapy for a minimum of 8 days.
  Arms: Standard antibiotic therapy

SUMMARY:
This study will enroll 460 subjects who have new pulmonary infiltrates during their ICU stay and who are at low risk of having pneumonia, as determined using the Clinical Pulmonary Infection Score (CPIS). The study is designed to determine whether 3 days of antibiotic treatment with meropenem (with or without coverage for MRSA) for ICU subjects diagnosed with new pulmonary infiltrates can reduce the emergence of anti-microbial-resistant organisms and the isolation of a potential pathogen compared to a standard course of antibiotic therapy (minimum of 8 days of therapy with antibiotics of the primary care team's choosing). Subjects will be randomly placed in either the meropenem group or standard antibiotic therapy group. The study will also examine whether short-course therapy reduces hospital length of stay and hospital cost, without having a negative effect on subject morbidity and mortality.

DETAILED DESCRIPTION:
Intensive care units (ICUs) are the most frequently identified source of nosocomial infections within the hospital, with infection rates and antimicrobial resistance rates significantly higher than in the general ward. In one study, antimicrobial use was reported to be 10 times higher in the ICU compared to antimicrobial use in the general ward. Although antibiotics are given for a variety of conditions, antibiotics prescribed for respiratory infections, suspected or proven, account for almost one-half of all antibiotic consumption in the ICU. Importantly, the use of antimicrobial agents has been identified as a critical risk factor in the emergence of resistant bacterial infections. By identifying and focusing on subsets of subjects who are unlikely to have infection and therefore unlikely to benefit from antibiotics, antibiotic use and the subsequent emergence of antimicrobial-resistant organisms could be limited. This is a Phase III, multi-center, randomized, open-label study designed to determine whether 3 days of antibiotic treatment with meropenem (with or without coverage for MRSA) for ICU subjects diagnosed with new pulmonary infiltrates can reduce the emergence of antimicrobial-resistant organisms and the isolation of a potential pathogen compared to a standard course of antibiotic therapy (minimum of 8 days of therapy with antibiotics of the primary care team's choosing). The primary objective of this study is to compare risk of resistant infection in the ICU by evaluating the difference in the incidence of either the emergence of antimicrobial-resistant bacteria or the isolation of a potential pathogen in ICU subjects who receive short-course empiric antibiotic therapy to ICU subjects who receive standard antibiotic therapy for the treatment of pulmonary infiltrates (with low likelihood of having pneumonia). Secondary objectives are to: 1) assess the mortality of subjects receiving short-course empiric antibiotic therapy compared to standard antibiotic therapy; 2) assess the ICU length of stay (LOS) in subjects receiving short-course empiric antibiotic therapy compared to standard antibiotic therapy; 3) assess the hospital LOS in subjects receiving short-course empiric antibiotic therapy compared to standard antibiotic therapy; 4) assess the costs of antibiotic therapy in subjects receiving short-course empiric antibiotic therapy compared to standard antibiotic therapy. The costs will be based on ICU LOS, hospital LOS, antibiotic treatment, and standard costs related to the treatment of infection-related adverse experiences; 5) assess the risk of clinically significant infection in subjects receiving short-course empiric antibiotic therapy compared to standard antibiotic therapy. This study will enroll 460 subjects who have new pulmonary infiltrates during their ICU stay and who are at low risk of having pneumonia, as determined using the Clinical Pulmonary Infection Score (CPIS).

ELIGIBILITY:
Inclusion Criteria:

1. Subject, or legal representative, has given written informed consent.
2. Subject has developed a new pulmonary infiltrate after ICU admission (confirmed by radiology).
3. Subject has been hospitalized at least three days.
4. CPIS </= 6.
5. 18 years of age or older.

Exclusion Criteria:

1. Burn patients.
2. Cystic fibrosis patients.
3. Bone marrow or solid organ transplant patients.
4. Neutropenia from any cause (absolute neutophil count (ANC) </= 500) or likely to become neutropenic within 7 days,
5. Known or suspected Human Immunodeficiency Virus (HIV) infection (HIV test is not required).
6. Suspected or proven extrapulmonary infection site requiring antibiotic therapy.
7. History of anaphylaxis to penicillin or cephalosporins.
8. History of anaphylaxis to meropenem (any component of the formulation) or other carbapenem (e.g., imipenem).
9. On systemic antibiotics for more than 7 consecutive days during the previous 30 days.
10. Received more than 2 doses of systemic antibiotics within the past 24 hours (other than those used for surgical prophylaxis),

9. Pregnant or lactating (Women of childbearing potential must have a negative serum or urine pregnancy test within the 7 days prior to the first dose of antibiotics).

10. Unlikely to survive past Day 7 of the study (as determined by the primary care team).

11. Previous enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Combined measure of either emergence of antimicrobial resistance or isolation of a potential pathogen detected in any positive clinical cultures that are deemed a clinically significant infection | Day 0 to day 28 (or hospital discharge, if earlier)

SECONDARY OUTCOMES:
ICU and Hospital length of stay (LOS) | Through Day 28 (or hospital discharge, if greater)
Health Economics: The costs will be based on ICU LOS, hospital LOS, antibiotic treatment, and standardized costs related to the treatment of infection-related adverse experiences. | Through Day 28 (or hospital dischange, if greater)
Any clinically significant infection, as determined by the subject's primary care team. | Through Day 28 (or hospital dischange, if greater)
Mortality rates at Days 14 and 28. | Days 14 and 28.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Christiana Care Health Services, Newark, Delaware
  - University of Miami, Miami, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Saint Patricks Hospital and Health Sciences Center, Missoula, Montana
  - Roswell Park Cancer Institute - Infectious Diseases, Buffalo, New York
  - Akron General Medical Center- Medicine, Akron, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - South Texas Veterans Health Care System, San Antonio, Texas